CLINICAL TRIAL: NCT07124793
Title: Phase II Study to Evaluate the Efficacy and Safety of IBI363 in Combination With IBI305 in Participants With Advanced Solid Tumors
Brief Title: A Study of IBI363 Combination Therapy in Participants With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363A203
Record Dates: First submitted 2025-08-07; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: EGFR Mutant NSCLC and Platinum Resistant Ovarian Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platinum resistant ovarian cancer (Experimental)
  Interventions: Drug: IBI363+IBI305
- EGFR mutant NSCLC cohort (Experimental)
  Interventions: Drug: IBI363+IBI305

INTERVENTIONS:
Drug: IBI363+IBI305 — Each treatment cycle lasts for 21 days (the first treatment cycle is 28 days). Subjects will receive IBI363 Q3W in combination with bevacizumab Q3W until 2 years of treatment, PD, intolerable toxicity, start of new anti-tumor treatment, withdrawal of informed consent, death, or study termination (whichever occurs first).

SUMMARY:
CIBI363A203, a Phase 2 study to evaluate the safety, tolerability and preliminary efficacy of IBI363 combined with IBI305 (a bevacizumab biosimilar) in participants with advanced malignancies conducted in China. Primary endpoint is objective response rate (ORR) per RECIST v1.1. Secondary endpoints include DoR, DCR, TTR, PFS, per RECIST v1.1, and OS; the incidence and severity of AEs, irAEs, SAEs, AESIs and their relationship to the investigational drug, and changes in vital signs, physical examination, and laboratory values before and after study treatment; PK, and immunogenicity of IBI363. The cohorts include: IBI363 and IBI305 combination therapy in participants with advanced EGFRmut NSCLC progressed after EGFR TKI and Platinum-based chemotherapy, and advanced platinum-resistant ovarian cancer (PROC). The anticipated enrollment for this study is approximately 60 participants with each cohort 30 participants, and actual enrollment may change with future amendments as cohorts are opened and closed based on evolving data.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be enrolled in the study:

1. Sign the written informed consent form and be able to comply with the visit arrangements and related procedures specified in the protocol.
2. Aged >= 18 years and <= 75 years, regardless of gender.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1.
4. Expected survival time >= 3 months.
5. Locally advanced or metastatic solid tumors confirmed by histology or cytology that are inoperable and cannot receive radical concurrent radiotherapy and chemotherapy:
6. Cohort A (EGFR-mutated NSCLC):

   * Histologically or cytologically confirmed unresectable locally advanced or metastatic non-small cell lung cancer;
   * Documented EGFR mutation (ex19del or L858R) detected in tumor tissue or blood samples;
   * Have progressed on or are intolerant to at least 1 prior line of approved EGFR TKI for metastatic or locally advanced NSCLC.T790M mutation requires 3rd generation TKI;
   * Patients with metastatic or locally advanced NSCLC who have shown progression or intolerance after at least 1 line of platinum-based chemotherapy;
   * Intolerance to or progression of the most recent line of anti-tumor therapy.
7. Cohort B (PROC):

   * Histologically or cytologically confirmed locally advanced unresectable or metastatic ovarian cancer, primary peritoneal cancer, or fallopian tube cancer;
   * Subjects with a documented breast cancer gene (BRCA) mutation (germline and/or somatic) must have been previously treated with a poly(ADP-ribose) polymerase (PARP) inhibitor;
   * For subjects with documented positive folate receptor-α (FRα) expression in tumor tissues, they should have previously received mirvetuximab soravtansine (MIRV) or ADC drugs with the same target, and have radiologically or pathologically confirmed PD;
   * Patients who have previously received ≥ 1 line of platinum-based chemotherapy and experienced progressive disease;

     * If you have only received 1 line of platinum-based chemotherapy, you must have received at least 4 cycles of platinum-based therapy, the best response is PR or CR, and disease progression occurs > 3 months and < 6 months after the last platinum-based chemotherapy;
     * If receiving 2 or more lines of platinum-based chemotherapy, must have had disease progression during or < 6 months after the last line of platinum-based chemotherapy Note: Disease progression is confirmed by imaging or pathology.
   * Must have received at least 1 line of prior systemic anti-cancer therapy:

     * Adjuvant ± neoadjuvant therapy is considered as first-line systemic anti-tumor treatment;
     * Maintenance therapy [e.g., bevacizumab and PARP inhibitors] as part of front-line anti-tumor treatment (the number of lines will not be counted separately);
     * For a change in treatment regimen, if the changed therapeutic drug is the same type of drug as the previous first-line treatment (for example, platinum, taxane, anthracycline, PARP inhibitor, etc. before and after the change), and there is no imaging disease progression before the change in therapeutic drug, the changed therapeutic regimen will be considered as part of the number of lines of treatment as before and will not be counted separately;
     * If the changed therapeutic drug is a different type of drug from the previous first-line treatment, or if radiographic disease progression occurs before the change of treatment, the number of lines needs to be calculated separately.
8. Adequate bone marrow and organ function:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; eosinophils < 1.5 × upper limit of normal (ULN); platelet count (PLT) ≥ 100 × 109/L; hemoglobin ≥ 9.0 g/dL; have not received treatment with erythropoietin (EPO), granulocyte-colony stimulating factor (G-CSF), or granulocyte-macrophage colony stimulating factor (GM-CSF) within 14 days prior to the first dose, and have not received blood transfusion (including red blood cell and platelet transfusion) within at least 14 days;
   * Liver function: total bilirubin ≤ 1.5 × ULN; AST and ALT ≤ 2.5 × ULN, without liver metastasis (if liver metastasis is present, ≤ 5 × ULN); albumin ≥ 3.0 g/dL (without albumin infusion within 14 days before the first dose);
   * Renal function: serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/min (using Cockcroft-Gault formula [Appendix 4]); and urine protein < 2+ or total 24-h urine protein < 1 g;
   * Coagulation function: International normalized ratio (INR) ≤ 1.5; activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN (subjects receiving anticoagulant therapy with coagulation function within the above range are allowed to be enrolled);
9. At least one measurable lesion according to RECIST v1.1.
10. For female subjects of childbearing age, a negative urine or serum pregnancy test within 7 days prior to receiving the first study drug administration. If the urine pregnancy test result is positive, a blood pregnancy test is required to be clearly negative or not pregnant;

Exclusion Criteria:

1. Cohort B (PROC) should not be enrolled if any of the following criteria is met based on histological or cytological findings:

   1. Documented sarcoma, mucinous carcinoma, undifferentiated carcinoma, or a combination thereof;
   2. Confirmed low-grade or borderline tumors, or contains the above components.
2. Previously received IL-2/IL-15 cytokine therapy. Except for the use of IL-2/IL-15 as an adjuvant component of adoptive cell therapy or as an immunomodulatory therapy for immunocompromised subjects.
3. Excluded medications and other treatments (subjects should not receive any of the following treatments):

   * Have received small-molecule targeted therapy or oral chemotherapy within 2 weeks or 5 half-lives (whichever is longer) before the first dose of the study drug; have received intravenous infusion of chemotherapy drugs within 3 weeks before the first dose of the study drug; have received Chinese herbal medicines with anti-tumor indications within 2 weeks before the first dose of the study drug;
   * Nitrosourea antineoplastic agents and mitomycin C within 6 weeks prior to the first dose of study drug;
   * Use of any antibody-based anti-tumor therapy within 4 weeks prior to the first dose of the study drug;
   * Participation in any medical device or other therapeutic interventional clinical trial within 2 weeks prior to the first dose of study drug;
   * Palliative radiotherapy within 2 weeks prior to the first dose of the investigational product, or radical radiotherapy within 4 weeks prior to the first dose;
   * Received adoptive cell therapy within 8 weeks prior to the first dose of study drug;
   * Use of live vaccines against infectious disease prophylaxis within 4 weeks prior to the first dose of study drug.
4. Active or untreated central nervous system metastasis (such as brain or leptomeningeal metastasis) confirmed by imaging assessment during screening or previous imaging assessment.

   * Subjects with asymptomatic brain metastases (i.e., no neurologically relevant symptoms, no corticosteroid treatment is required, and the diameter of metastatic lesions is ≤ 1.5 cm) may participate in this study.
   * Subjects whose symptoms of brain metastases are stable for ≥ 4 weeks after treatment and whose brain metastases do not increase in number or further increase after the end of treatment may participate in this study as long as they meet all of the following criteria:

     * Measurable lesions outside the central nervous system;
     * No metastases to meninges, midbrain, pons, medulla oblongata, or spinal cord; no multiple cerebellar metastases;
     * No compression of the aqueduct of the midbrain, no compression of the third or fourth ventricle, and no spinal cord compression;
     * Hormone therapy is discontinued 14 days prior to the first dose of the study drug.

   Note: Central nervous system lesions are not considered target lesions.
5. The tumor invades surrounding important tissue structures (such as mediastinal great vessels, superior vena cava, inferior vena cava, pericardium, heart, trachea, esophagus, etc.) or has the risk of gastrointestinal/respiratory fistula.
6. The subject has a history of significant toxicity related to immune checkpoint inhibitor administration and requires permanent discontinuation of the treatment.
7. Subjects with adverse reactions related to any previous anti-tumor treatment that have not recovered to Grade 0-1; except for persistent Grade 2 alopecia, peripheral neuropathy, hypomagnesemia, toxicities that are expected to be unrecoverable but stably controlled by the drug, and other conditions that the investigator considers to have no safety risk.
8. Have not recovered sufficiently from previous surgery, or have undergone any major surgery within 4 weeks prior to the first dose of the study drug.
9. Cardiovascular and cerebrovascular diseases with significant clinical significance, including:

   * Ventricular arrhythmia or other uncontrolled arrhythmias requiring medical intervention, such as antiarrhythmic drug therapy, etc.;
   * Severe conduction disorders (e.g., 3rd degree atrioventricular block);
   * HR-corrected QT interval (QTc interval, calculated using the Fridericia method [Appendix 5]) ≥ 480 ms;
   * Uncontrolled hypertension (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg) despite of standard treatment;
   * History of myocarditis;
   * Congestive heart failure currently requiring treatment;
   * Left ventricular ejection fraction (LVEF) < 50%;
   * Class III or IV cardiovascular disease according to New York Heart Association (NYHA) functional classification;
   * History of acute coronary syndrome (including myocardial infarction and unstable angina), coronary angioplasty or stenting within 6 months prior to the first dose of the study drug;
   * History of any arterial thromboembolic events within 6 months prior to the first dose of study treatment, including myocardial infarction, unstable angina, cerebrovascular accident, etc.
   * History of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolic event within 3 months prior to the first dose of study drug (thrombus or catheter-derived thrombus caused by an implanted venous port or superficial venous thrombosis is not considered a serious thromboembolism).
   * Known active seizures.
10. Subjects with interstitial pneumonia requiring steroid hormones or other treatments, or a history of other clinically significant lung diseases (such as pulmonary fibrosis, pneumoconiosis, interstitial lung disease, non-infectious pneumonia), or uncontrolled lung diseases (such as pulmonary fibrosis, severe radiation pneumonitis and acute lung injury) or suspected of having such diseases through imaging examinations during the screening period.
11. Allergic constitution, asthma, history of atopic dermatitis.
12. Pleural effusion, abdominal effusion or pericardial effusion requiring drainage or with obvious symptoms.
13. Active autoimmune diseases requiring systemic treatment (such as the use of disease-modifying drugs, corticosteroids or immunosuppressants) occurred within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments.
14. Have used immunosuppressive drugs within 14 days before the first study treatment, excluding intranasal and inhaled corticosteroids, or use systemic corticosteroids with a dose of less than 10 mg/day prednisone (or other corticosteroids with an equivalent dose to 10 mg/day prednisone), or use corticosteroids to prevent allergy to contrast agents.
15. Known allogeneic organ transplantation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through out the study (up to 2 years)

SECONDARY OUTCOMES:
disease control rate (DCR) | Through out the study (up to 2 years)
  To evaluate the preliminary antitumor activity of IBI363 plus bevacizumab.
duration of response (DoR) | Through out the study (up to 2 years)
  To evaluate the preliminary antitumor activity of IBI363 plus bevacizumab.
time to response (TTR) | Through out the study (up to 2 years)
  To evaluate the preliminary antitumor activity of IBI363 plus bevacizumab.
progression-free survival (PFS) | Through out the study (up to 2 years)
  To evaluate the preliminary antitumor activity of IBI363 plus bevacizumab.
Overall survival (OS) | Through out the study (an average of 2 years)
  To evaluate the preliminary antitumor activity of IBI363 plus bevacizumab.
Adverse Enent (AE) | Up to 90 days after the last administration
  AE is defined as an unexpected medical problem that happens during treatment with a drug or other therapy.
Treatment-Emergent AE (TEAE) | Up to 90 days after the last administration
  A TEAE will be defined as any new AE that begins, or any pre-existing condition that worsens in severity, after at least 1 dose of study treatment has been administered.
Immune-related AE (irAE) | Up to 90 days after the last administration
  irAE is defined as all grades of adverse drug reactions in clinical trials of anti-tumor drugs/therapies that are determined to be causally related to immune mechanisms.
Adverse Event of Special Interest (AESI) | Up to 90 days after the last administration
  AESI (Adverse Event of Special Interest) refers to adverse events that require special close monitoring to enhance the understanding of the investigational drug's safety. AESIs may be non-serious events.
Serious Adverse Event (SAE) | Through out the study (up to 2 years)
  An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is an important medical event that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before.
Plasma concentration (Cmax) of IBI363 | Up to 2 years
  PK parameters to be evaluated for IBI363 including maximum concentration (Cmax) will be determined when appropriate.
Area under the curve (AUC) of IBI363 | Up to 2 years
  PK parameters to be evaluated for IBI363 including area under the curve (AUC) will be determined when appropriate.
Half-life (T1/2) of IBI363 | Up to 2 years
  PK parameters to be evaluated for IBI363 including half-life (t1/2) will be determined when appropriate.
Clearance (CL) of IBI363 | Up to 2 years
  PK parameters to be evaluated for IBI363 including clearance (CL) will be determined when appropriate.
Volume of distribution (V) of IBI363 | Up to 2 years
  PK parameters to be evaluated for IBI363 including volume of distribution (V) will be determined when appropriate.
Immunogenicity of IBI363 | Up to 2 years
  Each subject will be tested for anti-drug (IBI363) antibody (ADA), and ADA-positive serum samples will continue to be tested for neutralizing antibodies (NAb).

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College HUST, Wuhan, Hubei, China